CLINICAL TRIAL: NCT04657393
Title: Prospective Comparison of Ventilation Patterns During Cardio-Pulmonary Resuscitation for Out-Of-Hospital Cardiac Arrest
Brief Title: Ventilation in Cardiac Arrest
Acronym: VICA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow inclusion
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VICA
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Cardio Respiratory Arrest; Cardiac Death; Ventilation Therapy; Complications; Apnea
Keywords: cardiopulmonary resuscitation; mechanical ventilation; Gas exchange
MeSH Terms: conditions — Heart Arrest; Death; Apnea | interventions — Respiration, Artificial

STUDY DESIGN:
Intervention Model Description: prospective, randomized, parallel study
Who Masked: Participant
Masking Description: randomizing the study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alternative Ventilation Rate (Active Comparator): ventilation is performed at 20 breaths/min
  Interventions: Procedure: mechanical ventilation
- Conventional Ventilation Rate (Active Comparator): ventilation is performed at 10 breaths/min
  Interventions: Procedure: mechanical ventilation

INTERVENTIONS:
Procedure: mechanical ventilation — change of ventilation frequency

SUMMARY:
Over the last decades, research in cardiopulmonary resuscitation was primarily focused on uninterrupted chest compressions to restore sufficient circulation. Ventilation during ongoing chest compressions was regarded as potentially deleterious and thus not given any major scientific focus. Current guidelines advise that ventilation be monitored by end-tidal CO2 and emphasize that hyperventilation be avoided. Recent findings from arterial blood gas analyses showed high levels of arterial pCO2, resulting in a frequent occurrence of hypercapnic acidosis, which may be caused by iatrogenic hypoventilation. Ventilation during ongoing chest compressions can be hard to achieve, as nearly every breath may be terminated by simultaneous chest compressions. In case of bag ventilation the applied tidal volumes have not yet been measured und mechanical ventilators so far were not able to ventilate during chest compressions, because pressure limit settings induced termination of inspiration.

The aim of this study is to provide patients with the best possible ventilation, even under ongoing chest compressions. Patients are ventilated with a new turbine-driven ventilator (Monnal T60, Air Liquide, France), which can deliver adequate tidal volumes within a very short inspiratory phase due to the inspiratory flow of > 200l/min. Thus, in deviation from the current recommendations, the ventilation rate can be doubled to 20/min, so that inspiration coincides with cardiac massage less often. The study compares effective ventilation volumes applied by two regimes, 10 breaths/min and 20/min.

DETAILED DESCRIPTION:
Restoration of circulation is undoubtedly the basis of success in cardiopulmonary resuscitation (CPR). Current guidelines on CPR require that hyperventilation be avoided during CPR. Blood gas analysis results from the "BABICA trial" demonstrate that more than 90% of patients have highly elevated levels of pCO2 and are acidotic, mainly due to hypercapnia. No hyperventilated or alkalotic patients were found during CPR. Furthermore, higher pO2 values were found to be associated with improved outcomes. Current recommendations to limit ventilation frequency to 10/min was also critically questioned in a recent study from Belgium, which did not show any positive effect of low respiration rate compared to higher ones, cut-off 10/min. There are currently no clinical trials addressing optimal tidal volumes or minute volumes during CPR.

A major obstacle to continuous measurement of respiratory minute volumes during CPR are ongoing chest compressions. In a retrospective study in which respiratory volumes were derived from bioimpedance curves, better outcomes were found in the group of more frequent ventilations. Common machine ventilators display set values, while expiratory volumes are averaged and may be overlaid by volume shifts of cardiac massage. In a recent study, investigators analyzed flow curves, where each breath can be evaluated individually and volumes can be derived correctly using dedicated software. We were able to test this method on a comparative study of three ventilators study on anatomical cadavers.

This study aims to detect whether a higher rate of ventilation using a turbine driven ventilator is able to provide higher breathing volumes during ongoing chest compressions in individuals suffering from out-of-hospital cardiac arrest (OHCA). Higher ventilation and oxygenation parameters as well as optimized acid-base-balance and increased rates of ROSC are expected.

Patient care (chest compressions, venous access, endotracheal intubation, application of drugs, defibrillation if necessary) is conducted according to current recommendation for Advanced Life Support (ALS) as issued by the European Resuscitation Council (ERC). Ventilation is performed at one of two patterns: the control group is ventilated at 10 breaths per minute, the intervention group is ventilated at 20 breaths per minute. Patterns are alternating according to calendar week. After successful endotracheal intubation mechanical ventilation is carried out using a turbine-driven ventilator (Monnal T60, AirLiquide, France). Ventilator settings are pre-set: respiratory frequency is set at 10/min or 20/min (see above), other ventilator parameters remain identical: Positive End-Expiratory Pressure (PEEP) 0 mmHg, FiO2 1,0, tidal volume 6ml/kg ideal body weight [men: 50+(0.91x(body length-152.4)), women: 45+(0.91y(body length-152.4))]. These calculations can be performed on the ventilator itself by entering patients' age, height and gender. Chest compressions are carried out without interruptions and without considerations regarding the respiratory cycle.

ELIGIBILITY:
Inclusion Criteria:

* out-of-hospital cardiac arrest (OHCA)
* cardio-pulmonary resuscitation (CPR) efforts
* endotracheal intubation

Exclusion Criteria:

* children and adolescents (age<18 years at inclusion)
* pregnant women
* previous documented lack of legal capacity
* previous documented refusal to participate in trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Minute ventilation | during ongoing chest compressions
  exspiratory ventilatory volume per minute
adequacy of ventilation - pH | during ongoing cardiopulmonary resuscitation
  Evaluation of ventilation success per using arterial blood gas analyses (pH)
adequacy of ventilation - paCO2 | during ongoing cardiopulmonary resuscitation
  Evaluation of ventilation success per using arterial blood gas analyses (paCO2)

SECONDARY OUTCOMES:
ROSC | during prehospital resuscitation efforts
  Return of Spontaneous Circulation

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prause, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Prause G, Zoidl P, Eichinger M, Eichlseder M, Orlob S, Ruhdorfer F, Honnef G, Metnitz PGH, Zajic P. Mechanical ventilation with ten versus twenty breaths per minute during cardio-pulmonary resuscitation for out-of-hospital cardiac arrest: A randomised controlled trial. Resuscitation. 2023 Jun;187:109765. doi: 10.1016/j.resuscitation.2023.109765. Epub 2023 Mar 15. PMID 36931453